CLINICAL TRIAL: NCT02441881
Title: A Double Blind Randomised Controlled Trial of Radiofrequency Thermo-ablation Treatments of Great Saphenous Varicose Veins: Venefit (Closurefast) vs. Radiofrequency Induced Thermal Therapy (RFITT) vs. Endovenous Radiofrequency (EVRF).
Brief Title: Trial of Radiofrequency Thermo-ablation Treatments of Great Saphenous Varicose Veins (3-RF Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Worcestershire Acute Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14/LO/1232
Record Dates: First submitted 2015-04-27; First posted 2015-05-12 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Varicose Veins
Keywords: Radiofrequency ablation; varicose veins; endothermal ablation; RFITT; Venefit
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Venefit (Active Comparator): Endovenous radiofrequency ablation device for truncal great saphenous vein ablation
  Interventions: Device: Venefit
- Radiofrequency Induced Thermal Therapy (Active Comparator): Endovenous radiofrequency ablation device for truncal great saphenous vein ablation
  Interventions: Device: Radiofrequency Induced Thermal Therapy
- Endovenous Radiofrequency (Active Comparator): Endovenous radiofrequency ablation device for truncal great saphenous vein ablation
  Interventions: Device: Endovenous Radiofrequency

INTERVENTIONS:
Device: Venefit — Endovenous radiofrequency device
  Other Names: Closurefast
  Arms: Venefit
Device: Radiofrequency Induced Thermal Therapy — Endovenous radiofrequency device
  Other Names: RFITT
  Arms: Radiofrequency Induced Thermal Therapy
Device: Endovenous Radiofrequency — Endovenous radiofrequency device
  Other Names: EVRF
  Arms: Endovenous Radiofrequency

SUMMARY:
A double blind randomised controlled trial of radiofrequency thermal ablation treatments of great saphenous varicose veins: Venefit (Closurefast), vs. Radiofrequency induced Thermal Therapy vs. Endovenous Radiofrequency.

Assessments by visual pain scores, duplex ablation and quality of life questionaires

DETAILED DESCRIPTION:
Purpose To establish which of the radiofrequency venous ablation modalities is most effective in preventing reflux in the treated segment of GSV six months following surgery.

Design Results of randomised trials and meta-analyses have shown that endovenous thermal ablation using radiofrequency ablation and laser are associated with improved recovery compared with conventional surgery on the GSV. Further, radiofrequency (Closurefast) has been showed to cause less pain and require less analgesic intake than laser. There are two other radiofrequency devices that have theoretical advantages over the Closurefast technique. All three procedures have been used in clinical practice (including at Worcestershire Royal Hospital). There has been no trial to date which has directly compared the outcomes of the three radiofrequency thermal ablation devices.

Recruitment Patients will be recruited from Worcestershire Acute Hospitals NHS Trust vascular surgical out-patient clinics. All patients will receive a duplex scan (Toshiba Viamo Ultrasound, Tokyo, Japan or Sonosite M-Turbo Bothell, Washington, USA) prior to entry into the trial to confirm their suitability for endovenous thermal ablation treatment. During this assessment patients will also have their CEAP (Clinical, Etiological, Anatomical, and Pathophysiological) classification of severity and aetiology of venous disease score recorded. If the patient consents to the trial they will be asked to fill in the disease specific Aberdeen Varicose Vein Questionnaire (AVVQ)and generic quality of life SF-36 and Euroquol (EQ-5D) questionnaires and have their Venous Clinical Severity Score (VCSS) calculated.

Patients will be recruited to the trial following an appropriate explanation of the study (see patient information / consent sheet). Randomisation will be performed by a random number generator (www.random.org).

Patients will be randomised to radiofrequency ablation either by Closurefast (Venefit, VNUS Medical Technologies, Inc., Sunnyvale, CA), the Radiofrequency induced Thermal Therapy (RFiTT, Olympus Surgical Technologies Europe, Hamburg, Germany) or EndoVenous Radiofrequency (EVRF, Medical Innovations, Bolton, United Kingdom). All treatments are already in use in Worcestershire.

Operation All treatments will be performed under local tumescent anaesthesia. Patients will receive thromboprophylaxis when indicated in line with the Hospital Trust's local thromboprophylaxis protocol. Procedures will be performed under duplex control (Sonosite M-Turbo, Bothell, Washington, USA) by an experienced vascular surgery Specialist Registrar or Consultant. The GSV will be catheterised percutaneously using a Seldinger technique at the level of the lowest point of reflux. The radiofrequency treatment catheter will be passed endoluminally to the level of the sapheno-femoral junction. Tumescent anaesthesia (50mg Prilocaine, 10mls 8.4% sodium bicarbonate in 1000mls 0.9% saline) will be injected in the peri-venous space in all patients (200 - 500ml). The position of the radiofrequency catheter will be confirmed just below the level of the sapheno-femoral junction prior to commencing the radiofrequency current and withdrawing the catheter to treat the vein in line with local practice. The Closurefast is withdrawn after a double treatment of the most proximal segment of the long saphenous vein and then segmentally thereafter, the RFiTT will be withdrawn continuously with retreatments, and the EVRF will be withdrawn in small stepwise movements (all as per the manufacturer's instructions for use). The volume of anaesthetic administered, length of vein treated and duration of the ablation will be recorded.

In line with current NICE guidance (CG168), where necessary, patients will undergo avulsions of local varicosities at the same time. The number of avulsions will be recorded in both groups. Perforating veins will not be directly treated. Treated legs will be dressed with dressing pads a full length bandage (coban, 3M United Kingdom plc, Bracknell, Berkshire, UK) and compression hosiery. Patients will be discharged on the day of surgery (day-case) with oral analgesia as required and will be given contact information should any adverse events arise.

Post-operative follow-up

i) First week Patients will be asked to keep a pain score for the first post-operative week. This is a simple 10cm visual analogue score. All patients will be invited back to clinic at two weeks for a duplex scan (blind assessment). During this visit the vascular team will assess any complications in the area of ablation including bruising (digital photographic record), wound infection, neuralgia, deep vein thrombosis and pulmonary embolus.

ii) Six months The primary endpoint of the study is an ablated GSV. Treatment failure will be defined as any segment of the treated trunk (> 2cm from the saphenofemoral junction) that is patent (compressible) and demonstrates reflux (>1 second) on duplex scanning.

A number of secondary outcome measures will be evaluated in the study:

Pain score/ analgesic requirements

Time to return to normal activity

Absence or recurrent varicose veins/return of symptoms

Quality Of Life (QoL): Disease specific (AVVQ) and generic (EQ5D & SF36) quality of life assessments will be compared at 1 weeks post treatment, 6 months and 12 months. The 1-week questionnaire will be given to the patient at discharge, whereas other QoL questionnaires will be sent to the patient. AVVQ is the most widely utilised disease specific QoL tool in venous disease and has been extensively validated. A score out of 100 points is calculated, with a higher score indicating more severe QoL impairment.

Other Markers Of Clinical Success: The Venous Clinical Severity Score (VCSS) will be assessed at 6 months. In addition, the incidence of complications related to the endovenous intervention as well as the presence of residual / recurrent varicose veins will also be assessed at 2 weeks.

Medium and longer-term endpoints (follow-up) will be performed at 2 years and 5 years. However, this is likely to be limited by the high rates (>20%) of drop-out reported in other studies.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic primary varicose veins of the great saphenous vein (GSV)
* Able to give informed consent to participate in the study after reading the patient information sheet
* Patients aged >18 years and < 80 years
* Ankle Brachial Pressure Index (ABPI) >/= 0.8

Exclusion Criteria:

* Unable to give informed consent
* Pregnancy (female participants of reproductive age will be eligible for inclusion in the study, subject to a negative pregnancy test prior to randomisation)
* Tortuous GSV not amenable to endovenous treatment
* Recurrent varicose veins (previous surgery)
* Presence of deep venous occlusive disease or other conditions precluding superficial venous intervention (at the discretion of the research team)
* Patients who are needle phobic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with 100% ablation of the previously treated vein segment | 6 months
  Duplex confirmed absence of recanalisation of the ablated

SECONDARY OUTCOMES:
Pain score on the visual scale | 7 days
  Percentage of patients scoring pain in each category for the three treatments
Quality of life measured by SF36, Euroqual 5D and Aberdeen varicose veins questionnaire | 12 months
  Quantitative and qualitative comparison of 3 trial populations

CONTACTS AND LOCATIONS:
Overall Officials: Isaac K Nyamekye, MD, FRCS, Principal Investigator — Worcestershire Acute Hospitals NHS Trust
Locations (1):
- Worcestershire Royal Hospital, Worcester, Worcestershire, United Kingdom

REFERENCES:
- [Derived] Nyamekye IK, Dattani N, Hayes W, Harding D, Holloway S, Newman J. A Randomised Controlled Trial Comparing Three Different Radiofrequency Technologies: Short-Term Results of the 3-RF Trial. Eur J Vasc Endovasc Surg. 2019 Sep;58(3):401-408. doi: 10.1016/j.ejvs.2019.01.033. Epub 2019 Jul 24. PMID 31351832
- [Derived] Gough MJ. Radiofrequency Venous Ablation: Not Simple and Not Always Effective! Eur J Vasc Endovasc Surg. 2019 Sep;58(3):409. doi: 10.1016/j.ejvs.2019.04.010. Epub 2019 May 21. No abstract available. PMID 31126836